CLINICAL TRIAL: NCT02979847
Title: Role of Epicardial Mapping and Ablation for Redo Procedure in Patients With Non-paroxysmal Atrial Fibrillation: a Prospective Randomized Trial
Brief Title: Epicardial Approach in Recurred Atrial Fibrillation
Acronym: EPIREAF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Korea University Anam Hospital (Other)
Responsible Party: Principal Investigator, Young-Hoon Kim, MD, Professor, Korea University Anam Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2016AN0127
Record Dates: First submitted 2016-09-11; First posted 2016-12-02 (Estimated); Last update posted 2020-11-17 (Actual); Status verified 2020-11

CONDITIONS: Persistent Atrial Fibrillation
Keywords: persistent atrial fibrillation; catheter ablation; epicardial mapping and ablation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Intervention Model Description: Randomized
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treated (Experimental): hybrid approach (epicardial and subsequent endocardial mappings and ablations)
  Interventions: Procedure: hybrid approach
- Control (Active Comparator): conventional endocardial approach
  Interventions: Procedure: conventional endocardial approach

INTERVENTIONS:
Procedure: hybrid approach — Before transseptal puncture, epicardial puncture is performed through subxyphoid approach. Atrial epicardial potentials are recorded using multi-electrode catheter, leading an activation map for atrial tachycardia and map for continuous fractionated atrial electrograms during atrial fibrillation. Endocardial potentials are also recorded in the same fashion. Procedural endpoint is a tachycardia termination or a noninducibility of tachycardia.
  Arms: Treated
Procedure: conventional endocardial approach — Atrial endocardial potentials are recorded using multi-electrode catheter, leading an activation map for atrial tachycardia and map for continuous fractionated atrial electrograms during atrial fibrillation. Procedural endpoint is a tachycardia termination or a noninducibility of tachycardia.
  Arms: Control

SUMMARY:
We aimed to assess the benefit of epicardial mapping and ablation in patients with recurred atrial tachyarrhythmias after single procedure for atrial fibrillation. We hypothesize that both endocardial and epicardial approach is superior to only endocardial approach with regards to clinical recurrence. Participants are randomized into a hybrid approach or an endocardial approach.

DETAILED DESCRIPTION:
Atrial electrical activity during atrial fibrillation depends on the distribution of myocardial tissue. Circumferential and longitudinal muscular bundles are multi-level crossing across the entire thickness of atrial wall. At radiofrequency catheter ablation for atrial fibrillation, transmural lesions are important to reduce the arrhythmogenic substrates and to prevent recurrence of scar-related atrial tachyarrhythmias.

Radiofrequency ablation applying electric current depends on impedance between patch and the tip electrode of a catheter. Increased impedance results in increased tissue heating, following an irreversible damage. However, overheating limits to create deep lesion formation because an increased impedance impedes the energy delivery to tissue. Furthermore, prolonged ablation time may result in severe complications, such as steam pop, cardiac perforation, and char formation. Therefore, both endocardial and epicardial ablations may be more effective to create a transmural lesion compared with only endocardial ablation.

Organized atrial tachycardia is common in patient who underwent ablation for atrial fibrillation. Activation mapping for atrial tachycardia is critical for ablating an isthmus. However, when the amplitude of endocardial potentials after previous ablations is decreased as system does not detect, summation of data from endocardium may give us wrong information about atrial tachycardia. Data from epicardial potential during tachycardia may be helpful to terminate a tachycardia.

We aimed to assess the benefit of epicardial mapping and ablation in patients with recurred atrial tachyarrhythmias after single procedure for atrial fibrillation. We hypothesize that both endocardial and epicardial approach is superior to only endocardial approach with regards to clinical recurrence. Participants are randomized into a hybrid approach or an endocardial approach.

ELIGIBILITY:
Inclusion Criteria:

* Patients with persistent AF (AF episode lasting > 7 days)
* Patients with symptomatic AF that is refractory to at least one antiarrhythmic medication
* Patients with recurrent arrhythmia after prior catheter ablation
* Patients undergoing a repeat ablation procedure for AF
* At least one episode of AF must have been documented by ECG, Holter, loop recorder, telemetry, trans telephonic monitoring (TTM), or implantable device within last 2 years of enrollment in this investigation
* Patients must be able and willing to provide written informed consent to participate in this investigation

Exclusion Criteria:

* Patients with permanent AF;
* Permanent AF will be defined as a sustained episode lasting more than 1 years and sinus rhythm never be observed .
* Patients for whom cardioversion or sinus rhythm will never be attempted/pursued;
* Patients with AF felt to be secondary to an obvious reversible cause
* Patients with contraindications to systemic anticoagulation with heparin or warfarin or a direct thrombin inhibitor;
* Moderate to severe valvular disease
* Patients who are pregnant. Pregnancy will be assessed by patients informing the physicians.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2016-06-29 (Actual); Primary Completion 2020-05-29 (Actual); Study Completion 2020-11-11 (Actual)

PRIMARY OUTCOMES:
Freedom from AF/AT recurrence | 12 months
  Freedom from sustained AF/AT recurrence Sustained AF/AT: sustained more than 30 sec documentation in clinical electrocardiography, Holter, event recorder

SECONDARY OUTCOMES:
Freedom from AF/AT recurrence without anti-arrhythmic drug use | 12 months
  Freedom from sustained AF/AT recurrence without anti-arrhythmic drug use
Freedom from AF recurrence | 12 months
  Freedom from sustained AF recurrence
Freedom from AT recurrence | 12 months
  Freedom from sustained AT recurrence
Procedure Time | Immediately after procedure
  From skin to skin
Fluoroscopic Time | Immediately after procedure
  Fluoroscopic Time
Ablation Time | Immediately after procedure
  Ablation Time
Procedure-related Acute Complications | Immediately after procedure
  Procedure-related Acute Complications
Procedure-related Subacute Complications | 3 months after procedure
  Procedure-related Subacute Complications

CONTACTS AND LOCATIONS:
Overall Officials: Young-Hoon Kim, MD, PhD, Principal Investigator — Korea University
Locations (1):
- Korea University Medical Center Anam hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No
The individual participant data is not available to share with other researchers.

REFERENCES:
- [Result] Eckstein J, Zeemering S, Linz D, Maesen B, Verheule S, van Hunnik A, Crijns H, Allessie MA, Schotten U. Transmural conduction is the predominant mechanism of breakthrough during atrial fibrillation: evidence from simultaneous endo-epicardial high-density activation mapping. Circ Arrhythm Electrophysiol. 2013 Apr;6(2):334-41. doi: 10.1161/CIRCEP.113.000342. Epub 2013 Mar 19. PMID 23512204
- [Result] Lee G, Kumar S, Teh A, Madry A, Spence S, Larobina M, Goldblatt J, Brown R, Atkinson V, Moten S, Morton JB, Sanders P, Kistler PM, Kalman JM. Epicardial wave mapping in human long-lasting persistent atrial fibrillation: transient rotational circuits, complex wavefronts, and disorganized activity. Eur Heart J. 2014 Jan;35(2):86-97. doi: 10.1093/eurheartj/eht267. Epub 2013 Aug 8. PMID 23935092
- [Result] Lee G, Spence S, Teh A, Goldblatt J, Larobina M, Atkinson V, Brown R, Morton JB, Sanders P, Kistler PM, Kalman JM. High-density epicardial mapping of the pulmonary vein-left atrial junction in humans: insights into mechanisms of pulmonary vein arrhythmogenesis. Heart Rhythm. 2012 Feb;9(2):258-64. doi: 10.1016/j.hrthm.2011.09.010. Epub 2011 Sep 9. PMID 21907170
- [Result] Pak HN, Hwang C, Lim HE, Kim JS, Kim YH. Hybrid epicardial and endocardial ablation of persistent or permanent atrial fibrillation: a new approach for difficult cases. J Cardiovasc Electrophysiol. 2007 Sep;18(9):917-23. doi: 10.1111/j.1540-8167.2007.00882.x. Epub 2007 Jun 16. PMID 17573836
- [Result] Verheule S, Tuyls E, Gharaviri A, Hulsmans S, van Hunnik A, Kuiper M, Serroyen J, Zeemering S, Kuijpers NH, Schotten U. Loss of continuity in the thin epicardial layer because of endomysial fibrosis increases the complexity of atrial fibrillatory conduction. Circ Arrhythm Electrophysiol. 2013 Feb;6(1):202-11. doi: 10.1161/CIRCEP.112.975144. Epub 2013 Feb 6. PMID 23390124
- [Result] Eckstein J, Schotten U. Rotors and breakthroughs as three-dimensional perpetuators of atrial fibrillation. Cardiovasc Res. 2012 Apr 1;94(1):8-9. doi: 10.1093/cvr/cvs093. Epub 2012 Feb 13. No abstract available. PMID 22331500